CLINICAL TRIAL: NCT06017323
Title: Phase I Study of Proglumide With Gemcitabine and Nab-Paclitaxel in Patients With Metastatic Pancreatic DuctalAdenocarcinoma
Brief Title: Proglumide With Gemcitabine and Nab-Paclitaxel in PatientsWith Metastatic Pancreatic Ductal Adenocarcinoma
Acronym: ProglumidePanc
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: STUDY00006987
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001899
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Proglumide; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Level 1:Proglumide TID with Gemcitabine and Nab-Paclitaxel (Experimental): Proglumide given three times a day with gemcitabine and nab-paclitaxel
  Interventions: Drug: Gemcitabine; Drug: Nab paclitaxel; Drug: Proglumide Dose level 1
- Dose Level 2:Proglumide BID with Gemcitabine and Nab-Paclitaxel (Experimental): Proglumide given two times a day with gemcitabine and nab-paclitaxel
  Interventions: Drug: Gemcitabine; Drug: Nab paclitaxel; Drug: Proglumide Dose level 2

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2 IV given days 1, 8, and 15every 28 days (1 cycle)
  Other Names: Gemzar
Drug: Nab paclitaxel — 125 mg/m2 given days 1, 8, and 15every 28 days (1 cycle)
Drug: Proglumide Dose level 1 — Daily dose of 1200 mg orally given as400 mg orally (PO), three times a day(TID) (dose level 1)
  Arms: Dose Level 1:Proglumide TID with Gemcitabine and Nab-Paclitaxel
Drug: Proglumide Dose level 2 — Daily dose of 1600 mg orally given as800 mg orally (PO) twice a day (BID)(dose level 2).
  Arms: Dose Level 2:Proglumide BID with Gemcitabine and Nab-Paclitaxel

SUMMARY:
This is a Phase I open labelled study to treat patients with metastatic pancreatic cancer with combination therapy using standard of care first line therapy with gemcitabine and nab-paclitaxel given days 1, 8, and 15 every 28 days, and proglumide. This is a phase 1 study with 3+3 design, enrolling3-12 patients over 2 planned dose levels of proglumide(maximum 6 patients per dose level). Proglumide will be tested at the daily dose of 1200 mg orally (PO) given as 400mg three times daily (TID) (dose level 1) or 1600 mg orally(PO) given as 800 mg twice a day (BID) (dose level 2). All cycles are 28 days. Patients will be monitored for safety and toxicity by laboratory blood testing and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (e.g., HIPAA in the USA) obtained from the patient prior to performing any protocol-related procedures, including screening evaluations
2. Age > 18 years at time of study entry.
3. Adequate normal organ and marrow function as defined below:

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) > 1500 permm3
   * Platelet count ≥100,000 per mm3)
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).
   * Aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤2.5 x ULN of normal unless liver metastases are present, in which case it must be ≤5x ULN
   * Creatinine clearance (CL) >60 mL/min using the Cockcroft-Gault formula.
4. Evidence of post-menopausal status or negative urine or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   -Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments, or if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization(bilateral oophorectomy or hysterectomy).
5. Patients must have measurable disease by RECIST v1.1 and disease amenable to serial biopsy.
6. Subjects may not have received prior therapy with Gemcitabine (GEM)/Nab-paclitaxel (NAB-P).
7. Patients must have metastatic pancreatic ductal adenocarcinoma with adenocarcinoma as the dominant histology (biopsy-proven, primary tumor biopsy is acceptable for eligibility)
8. No prior systemic treatment for metastatic disease(neoadjuvant/adjuvant therapy is allowable but could not contain GEM or NAB-P).
9. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Subjects with a concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer, or localized prostate cancer following definitive therapy.
2. Subjects with uncontrolled cardiovascular diseases(congestive heart failure, symptoms of coronary artery disease, cardiac arrhythmias) or who have suffered a myocardial infarction in the preceding 6months.
3. Blood anticoagulation that cannot be safely stopped for biopsy.
4. Subjects with poorly controlled medical conditions including asthma, chronic obstructive pulmonary disease, diabetes, seizure disorders, hepatic or renal failure.
5. Pregnant or nursing women.
6. Men or women of childbearing potential who are unwilling to employ adequate contraception(condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence) prior to study entry, for the duration of study participation, and for 6 months thereafter.
7. Any concurrent chemotherapy, Investigational Product (IP), biologic, or hormonal therapy for cancer treatment.
8. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
9. History of allogenic organ transplantation.
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea or inability to digest and absorb pills, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring Adverse Events (AEs) or compromise the ability of the patient to give written informed consent
11. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and Tuberculosis (TB) testing in line with local practice), hepatitis B (HBV) (known positive HBV surface antigen (HBsAg) result), hepatitis C (HCV), or human immunodeficiency virus (positive HIV 1/2 antibodies).

    * Patients with a past or resolved HBV infection(defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.
    * Patients positive for hepatitis C (HCV)antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
    * Testing for tuberculosis, hepatitis B and C and HIV is not a requirement for screening for the clinical trial.
12. Receipt of live attenuated vaccine within 30 days prior to the first dose of investigational drug. Note: Patients, if enrolled, should not receive live vaccine while receiving IP and up to 30 days after the last dose of IP.
13. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of proglumide therapy.
14. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
15. Patient is unable to swallow pills or has a malabsorption syndrome that would not enable the patient to properly absorb proglumide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proglumide Recommended Phase II dose and schedule (RP2D) | 2 years
  Determination of the recommended phase II dose and schedule (RP2D) of proglumide in combination with gemcitabine and nab-paclitaxel in patients with metastatic pancreatic ductal adenocarcinoma

SECONDARY OUTCOMES:
Overall survival (OS) | through 2 years after end of treatment
  median overall survival will be estimated using Kaplan-Meier curves.
Progression-free survival | 2 years
  median progression free survival will be estimated using Kaplan-Meier curves.
Objective response rate by RECIST v. 1.1 | 2 years
  Every 8 weeks (± 7 days) radiographic imaging (CT or MRI) will be done to assess tumor burden according to RECIST v. 1.1
Change in tumor marker (CA19-9) | 2 years
  Maximum percent decrease in CA19-9 will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin WE, MD, Principal Investigator — Georgetown University
Locations (1):
- Lombardi Comprehensive Cancer Center, Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No